CLINICAL TRIAL: NCT00668954
Title: Antioxidant Effects of Pomegranate Juice Versus Placebo in Adults With Type 2 Diabetes Mellitus Following a Glucose Load
Brief Title: Antioxidant Effects of Pomegranate Juice Versus Placebo in Adults With Type 2 Diabetes Mellitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: POM Wonderful LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 07-0878
Record Dates: First submitted 2008-04-25; First posted 2008-04-29 (Estimated); Last update posted 2015-07-31 (Estimated); Status verified 2015-07

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Diabetes; Pomegranate; Biomarkers; Antioxidant
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pomegranate Juice (Active Comparator)
  Interventions: Dietary Supplement: Pomegranate Juice
- Placebo Juice (non-Pomegranate) (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo Juice

INTERVENTIONS:
Dietary Supplement: Pomegranate Juice — Group A drinks 8 oz. pomegranate juice/day for 12 weeks
  Arms: Pomegranate Juice
Dietary Supplement: Placebo Juice — Group B drinks 8 oz. placebo juice/day for 12 weeks
  Arms: Placebo Juice (non-Pomegranate)

SUMMARY:
This is a research study designed to look at how pomegranate juice (or a placebo juice) affects the body through the measurement of specific biomarkers, which are indicators of health.

DETAILED DESCRIPTION:
This research study will evaluate how pomegranate juice (or a placebo juice) affects the body. Participants will be asked to drink 8 oz. of juice daily for 12 weeks. Biomarkers, which are indicators of health, will be measured throughout the study. They are present in blood and urine. The placebo is a juice that is not made from pomegranates, but resembles pomegranate juice in color and taste. Eating pomegranates has been shown to have a positive impact on certain biomarkers. Recent studies have shown that biomarkers can be indicators of general health. The investigators want to know if drinking pomegranate juice daily for 12 weeks is effective at improving a variety of biomarkers in diabetic adults.

ELIGIBILITY:
Inclusion Criteria:

* Able to speak and read English
* Have a diagnosis of Type II Diabetes Mellitus and currently being treated with oral medication
* Have an HbA1C level ≤9.0% at Screening
* Have an hsCRP level ≥ 1.0 at Screening
* 35 - 70 years old (inclusive)
* Non-smokers
* Willing to maintain his/her normal activity and eating patterns for the duration of the study
* Willing to maintain his/her normal diet for the duration of the study but avoid anti-oxidant rich foods and pomegranate juice (other than what is dispensed to them)

Exclusion Criteria:

* Allergy to pomegranates
* Currently using insulin
* Currently taking steroidal drugs
* HIV positive or AIDS
* Chronic infectious disease
* Recent (within 2 weeks of screening) cold/flu, inflammatory illness, or flare-up of gout
* Cancer treated within the past two years
* Participation in a therapeutic research study within 30 days of baseline
* Women who are pregnant, lactating, or planning to become pregnant during the study period

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2008-04; Primary Completion 2009-04 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Percent change of oxidant stress and lipid oxidation | baseline, week 6, week 12

SECONDARY OUTCOMES:
HbA1c | baseline, week 6, week 12
High Sensitivity C-reactive protein HsCRP | baseline, week 6, week 12

CONTACTS AND LOCATIONS:
Overall Officials: James O. Hill, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Denver Center for Human Nutrition, Denver, Colorado, United States